CLINICAL TRIAL: NCT05659914
Title: Olaparib and Durvalumab (MEDI4736) in Patients with Metastatic Pancreatic Cancer and DNA Damage Repair Genes Alterations
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Cooperative Group for the Treatment of Digestive Tumours (TTD) (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TTD-20-04; 2020-004859-32 (EudraCT Number)
Record Dates: First submitted 2022-11-22; First posted 2022-12-21 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: Metastatic Pancreatic Cancer; DDR genes; durvalumab; olaparib
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- olaparib +durvalumab (Experimental): olaparib+durvalumab
  Interventions: Drug: olaparib+durvalumab

INTERVENTIONS:
Drug: olaparib+durvalumab — olaparib: 300 mg tablets taken orally twice daily and durvalumab: 1500 mg via IV infusion q4w

SUMMARY:
Patients with metastatic pancreatic cancer and germline mutation in BRCA have benefit of therapy with PARP inhibitors. In addition, some studies have demonstrated that PDL-1 inhibitors synergize therapeutically with PARP inhibitors in tumours with homologous repair deficiency.

Our hypothesis is that those patients with alterations in DNA damage repair genes (somatic and germline BRCA1, BRCA2, PALB2, RAD51C, RAD51D and other functional DDR genes) and who have benefit from platinum based therapy in first line might obtain an increased therapeutic effect with the combination of olaparib and durvalumab.

This is an open-label, single-arm, multicentric phase II clinical trial of a combination of durvalumab and olaparib in patients with metastatic pancreatic cancer with alterations in DDR genes, who have had benefit with platinum-based chemotherapy in first line setting. The primary objective is to investigate the efficacy of this combination in terms of ORR.

Patients will be eligible for the study based on alterations in a panel of specific DDR genes including BRCA1, BRCA2, PALB2, RAD51C, RAD51D and other DDR genes, as determined by a local assay according to local practice or by the central laboratory (if local assay is not available).

ELIGIBILITY:
Inclusion Criteria:

Pre-screening Inclusion Criteria (not required for patients with alterations in DDR genes determined by local practice)

Subjects will be eligible for inclusion in pre-screening for the study only if all of the following criteria apply:

1. Males and females ≥18 years of age (at the time consent is obtained).
2. Written informed consent provided.
3. Performance Status score of 0 or 1 according to the Eastern Cooperative Oncology Group (ECOG) scale.
4. Subject must have archival tumour tissue available for central laboratory testing of alterations in DDR genes or willing to undergo a fresh tumour biopsy.
5. Histologically or cytologically confirmed adenocarcinoma of the pancreas. 5.1.2 Screening Inclusion Criteria

   Patients are eligible to be included in the study only if all of the following inclusion criteria and none of the exclusion criteria apply:
6. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Provision of signed and dated, written informed consent form prior to any mandatory study specific procedures, sampling, and analyses.
7. Male or female patients 18 years of age or older, at the time of signing the ICF.
8. Histologically or cytologically confirmed metastatic adenocarcinoma of the pancreas with alterations in DNA damage repair genes.
9. Presence of alterations in DDR genes in tumour tissue previously determined by a local assay at any time prior to Screening or by the central laboratory.
10. Patients must have received a minimum of 1 line of chemotherapy for advanced or metastatic disease and a maximum of 2 lines. Patients who have received adjuvant treatment and have recurrence within 6 months of completion of the adjuvant or neoadjuvant treatment, is counted as first line chemotherapy.
11. Patients must have received platinum-based chemotherapy and must have benefit of it and not progressed while on platinum. Benefit is defined as partial or complete response or PFS ≥ 6 months.
12. Patients must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below:

    * Haemoglobin ≥ 10.0 g/dL with no blood transfusion in the past 28 days.
    * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L.
    * Platelet count ≥ 100 x 109/L.
    * Total serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN).
    * Aspartate aminotransferase (AST) (Serum Glutamic Oxaloacetic Transaminase (SGOT)) / Alanine aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase (SGPT)) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present in which case they must be ≤ 5x ULN.
    * International normalized ratio (INR) ≤ 1.5 x ULN
    * Serum creatinine ≤ 1.5 x ULN
    * Total bilirubin ≤ 1.5 x ULN
    * Albumin >3g/dL
    * Measured creatinine clearance (CL) >51 mL/min or Calculated creatinine CL>51 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

    Males:

    Creatinine CL (mL/min) = Weight (kg) x (140 - Age) 72 x serum creatinine (mg/dL)

    Females:

    Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85 72 x serum creatinine (mg/dL)
13. Body weight >30 kg
14. ECOG performance status 0-1 within 14 days before enrolment (Appendix A).
15. Measurable disease as defined by RECIST version 1.1 guidelines.
16. Patients must have a life expectancy ≥ 16 weeks.
17. Postmenopausal or evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 7 days of study treatment.

    Postmenopausal is defined as:
    * Amenorrhoeic for 1 year or more following cessation of exogenous hormonal treatments.
    * Luteinizing hormone (LH) and Follicle stimulating hormone (FSH) levels in the post-menopausal range for women under 50.
    * radiation-induced oophorectomy with last menses >1 year ago.
    * chemotherapy-induced menopause with >1 year interval since last menses.
    * surgical sterilisation (bilateral oophorectomy or hysterectomy). Women who are of childbearing potential and sexually active must agree to the use of 1 highly effective form of contraception (see 5.3.1), and their partners must use a male condom, or they must totally/truly abstain from any form of sexual intercourse (see 5.3.1), throughout their participation in the study and for at least 3 months after last dose of study drug(s).
18. Male patients must use a condom during treatment and for 3 months after the last dose of study drug when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Female partners of male patients should also use a highly effective form of contraception (see 5.3.1) if they are of childbearing potential. Male patients should not donate sperm throughout the period of taking study drug and for 3 months following the last dose of study drug.
19. Resolution of all toxic effects of prior treatments except alopecia to Grade 0 or 1 by NCI CTCAE version 5.0.
20. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures.

Exclusion Criteria:

1. Other malignancy unless curatively treated with no evidence of disease for ≥5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), Stage 1, grade 1 endometrial carcinoma.
2. Uncontrolled, clinically significant, symptomatic cardiovascular disease within 6 months before enrolment, including myocardial infarction, unstable angina, grade 2 or greater peripheral vascular disease, cerebrovascular accident, transient ischemic attack, congestive heart failure, or arrhythmias not controlled by outpatient medication.
3. Resting ECG indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (e.g., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QTcF prolongation >500 ms, electrolyte disturbances, etc.), or patients with congenital long QT syndrome.
4. Persistent toxicities (>Common Terminology Criteria for Adverse Event (CTCAE) grade 2) caused by previous cancer therapy, excluding alopecia.
5. Patients with myelodysplastic syndrome/acute myeloid leukaemia or with features suggestive of MDS/AML.
6. Patients with symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days.
7. Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent.
8. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
9. Patients with an active infection.
10. Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV)
11. Patients with known active hepatitis (i.e., Hepatitis B or C).

    * Active hepatitis B virus (HBV) is defined by a known positive HBV surface antigen (HBsAg) result. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody and absence of HBsAg) are eligible.
    * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
12. Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent:

    * Participants with type 1 diabetes, vitiligo, alopecia, psoriasis, hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible.
    * Participants requiring hormone replacement with corticosteroids are eligible if the steroids are administered only for the purpose of hormonal replacement and at doses ≤ 10 mg of prednisone or equivalent per day.
13. Any pre-existing medical condition of sufficient severity to prevent full compliance with the study.
14. Have received previously treatment with PARP inhibitors or PDL-1 inhibitors (including durvalumab)
15. Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 3 weeks prior to study treatment
16. Concomitant chemotherapy, hormonal therapy, immunotherapy, or any other form of cancer treatment.
17. Concomitant use of known strong CYP3A inhibitors (e.g. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks.
18. Concomitant use of known strong (e.g. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort ) or moderate CYP3A inducers (e.g. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
19. Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
20. Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).
21. Concurrent treatment or treatment within 4 weeks of study entry with any other investigational agent.
22. Patients with a known hypersensitivity to olaparib, durvalumab or any of the excipients of the product.
23. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
24. Female patients who are lactating and breastfeeding or have a positive pregnancy test during the Screening Period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-11-28 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Baseline through the end of the study (up 42 months)
  ORR defined as the percentage of patients with an investigator-assessed complete (CR) or partial response (PR) according to Response Evaluation Criteria in Solid tumours (RECIST) v1.1.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Baseline through the end of the study (up 42 months)
  PFS defined as the time from initial date of study treatment to the date of objective disease progression according to RECIST 1.1 criteria or death (due to any cause), whichever occurs first
Overall survival (OS) | 42 months
  OS defined as the time from the initial date of the study treatment to the date of death (due to any cause), with patients alive or lost to follow-up at the analysis data cut-off date censored at their last contact date.
Duration of response (DoR) | Baseline through the end of the study (up 42 months)
  DoR defined as time from first objective response to disease progression per RECIST 1.1 criteria or death (due to any cause). For patients with response who have not progressed or died at last observation
Disease control rate (DCR) | Baseline through the end of the study (up 42 months)
  DCR defined as the percentage of patients who achieve complete response, partial response or stable disease.
Incidence and severity of AEs CTCAE v5 criteria | Baseline through the end of the study (up 42 months)
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0 and serious Adverse Events. Change From Baseline to the end of treatment in abnormal vital signs, abnormal ECG results and evaluation of laboratory parameters

OTHER OUTCOMES:
To characterize the immune microenvironment of this tumours and biomarkers of HRD status, and RAD51 status in tumour tissue samples and blood samples | Tumour tissue samples: at baseline and at progression and blood samples at baseline, on treatment and at progression
  To be assessed by Next-Generation Sequencing (NGS) analysis

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Macarulla, MD, Principal Investigator — Vall d'Hebron University Hospital
Locations (3):
- Spain (3):
  - Complejo Hospitalario Universitario La Coruña, A Coruña
  - Hospital Universitari Vall d´Hebron, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander